CLINICAL TRIAL: NCT03817385
Title: Effect of Repetitive Transcranial Magnetic Stimulation (rTMS) and Robotic Gait Training on Lower-extremity Function and Gait in Patients With Stroke
Brief Title: rTMS and Robotic Gait Training in Patients With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Ta-Sen Wei,MD, Director, Physical Medical and Rehabilitation, Principal Investigator, Clinical Professor, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCH-160102
Record Dates: First submitted 2018-12-28; First posted 2019-01-25 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Stroke
Keywords: Transcranial magnetic stimulation; Robotic gait training; Gait; Spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- repetitive TMS (Transcranial Magnetic Stimulation) (Experimental): rTMS and physical / occupational therapy
  Interventions: Device: repetitive TMS
- robotic GT (Gait Training) (Experimental): robotic gait training for 20 times and physical / occupational therapy
  Interventions: Device: robotic GT
- traditional rehabilitation (No Intervention): patient only received traditional rehabilitation program

INTERVENTIONS:
Device: repetitive TMS — rTMS x 10 times
  Arms: repetitive TMS (Transcranial Magnetic Stimulation)
Device: robotic GT — robotic gait training for 20 times
  Arms: robotic GT (Gait Training)

SUMMARY:
Patients with stroke have demonstrated abnormal muscle tone and postural control ability which affect their ambulation, activity of daily living and confident. Nowadays, utilizing repetitive transcranial magnetic stimulation (rTMS) and robotic machines to assist walking training for stroke patients has been applied to clinic widely. While less studies have compared intervention efficacy for stroke patients between rTMS and robotic training. This study aimed to compare effect of rTMS and robotic training for lower-extremity function and gait in stroke patients.

DETAILED DESCRIPTION:
This study will include subjects occurring stroke within 3 months. All groups will receive traditional rehabilitation. The subjects will be allocated randomly in three groups which are traditional rehabilitation (Group A), robotic training (Group B), and rTMS (Group C) respectively, with 35 people per group. The group B will be intervened 5 times per week and the group C will receive 10 times rTMS intervention during 4 weeks. At post-intervention and eighth weeks after intervention, basic examination will be executed including basic information, history, Mini-mental State examination, Short -Form 36, Modified Ashworth Scale, Fugl-Meyer assessment, static and dynamic motion examination, ultrasound assessment and examination of cardiorespiratory. Two-way mixed ANOVA will be used to analyze the differences of three groups and times.

ELIGIBILITY:
Inclusion Criteria:

* first-time onset of stroke
* reaching 20 years old and having clinical CT and MRI diagnosis of stroke
* hemiparesis with sitting ability after onset 3 months

Exclusion Criteria:

* Brunnstrom stage over grade V
* Combined other neurological diseases (epilepsy, polyneuropathy, Meniere's disease, vestibular neuritis, Parkinson's disease, dementia, spinocerebellar ataxia)
* lower extremity disease, included joint contracture, high muscle tone(MAS more than 3), L/E fracture, Joint replacement, long-term osteoarthritis pain
* unstable vital sign
* can't coordinate or Sign consent plan form

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Change of walking speed | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  walk 6m to measure the time spent, patients can walk with foot orthosis and assistive devices
Change of postural sway displacement | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  Use computerized dynography to measure the postural sway displacement (mm)
Change of postural sway velocity | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  Use computerized dynography to measure the postural sway velocity (mm/s)
Change of postural sway area | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  computerized dynography to measure the postural sway area (mm^2)
Change of step time | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  Use computerized dynography to measure spatial gait parameter: step time (ms)
Change of stance time | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  Use computerized dynography to measure spatial gait parameter: stance time (ms)
Change of swing time | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  Use computerized dynography to measure spatial gait parameter: swing time (ms)
Change of single support time | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  Use computerized dynography to measure spatial gait parameter: single support time (ms)
Change of double support time | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  Use computerized dynography to measure spatial gait parameter: double support time (ms)
Change of step length | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  Use computerized dynography to measure spatial gait parameter: step distance (mm)
Change of stance length | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  Use computerized dynography to measure spatial gait parameter: stance distance (mm)
Change of amplitude of Muscle activity | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  use electromyography to measure the muscles activity in microvolts (uv) included quadriceps, hamstrings, tibialis anterior, gastrocnemius during subject walking in self selected speed in 6 meters.
Change of Functional Independence Measure (FIM) | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  FIM™ is comprised of 18 items, grouped into 2 subscales - motor and cognition.
  The motor subscale includes:
  Eating Grooming Bathing Dressing, upper body Dressing, lower body Toileting Bladder management Bowel management Transfers - bed/chair/wheelchair Transfers - toilet Transfers - bath/shower Walk/wheelchair Stairs
  The cognition subscale includes:
  Comprehension Expression Social interaction Problem solving Memory Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item.
  The total score for the FIM motor subscale will be a value between 13 and 91. The total score for the FIM cognition subscale will be a value between 5 and 35.
  The total score for the FIM instrument will be a value between 18 and 126.
Change of international Quality of Life Assessment Short Form -36 (SF-36) | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  including 8 health concepts: (1) physical functioning, (2) role limitations because of physical health problems; (3) bodily pain, (4) social functioning, (5) general mental health (psychological distress and psychological wellbeing), (6) role limitations because of emotional problems, (7) vitality (energy/fatigue), (8) general health perceptions.
  Scoring: answers to each question are scored which are then summed and transformed to a 0 - 100 scale.

SECONDARY OUTCOMES:
Change of concentration of Serum albumin | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  The concentration of Serum albumin in the blood test. Albumin is the most important contributor to the maintenance of plasma colloid oncotic pressure; deficiency results in edema.because of physical health problems; (3) bodily pain, (4) social functioning, (5) general mental health (psychological distress and psychological wellbeing), (6) role limitations because of emotional problems, (7) vitality (energy/fatigue), (8) general health perceptions.
  Scoring: answers to each question are scored which are then summed and transformed to a 0 - 100 scale.
Change of concentration of Hemoglobin (Hb) | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  The concentration of Hb in the blood test.
Change of concentration of Glucose | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  The concentration of Glucose in the blood test. The Spot glucose measurement in epidermal interstitial fluid appears to be a promising alternative to capillary blood glucose estimation
Change of concentration of Cholesterol | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  The concentration of Cholesterol in the blood test.
Change of concentration of Triglyceride | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  The concentration of Triglyceride in the blood test.
Change of Berg balance test (BBS) | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  Including 14 items which are scored on a 5 points scale (0-4). The degree of success in achieving each task is given a score of zero (unable) to four (independent), and the final measure is the sum of all of the scores.
  The item scores are summed, minimum score =0, maximum score = 56
Change of Fugl-Meyer Assessment (FMA) | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  Items are scored on a 3-point ordinal scale (0 = cannot perform; 1 = performs partially; 2 = performs fully) Maximum Score = 226 points The 5 domains assessed include, Motor function (Upper extremity maximum score = 66; Lower extremity maximum score = 34), Sensory function (maximum score = 24), Balance (maximum score = 14), Joint range of motion (maximum score = 44), Joint pain (maximum score = 44)
Change of Body Mass Index (BMI) | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  (body weight) kg/(height) m*(height)m
Change of Mini-mental state examination (MMSE) | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  It is an 11-question measure that tests five areas of cognitive function:
  orientation, registration, attention and calculation, recall, and language. The maximum score is 30. A score of 23 or lower is indicative of cognitive impairment.
Change of Modified Ashworth scale (MAS) | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  measures resistance during passive soft-tissue stretching, the score is ranged from 0-4 0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of motion (ROM)
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
Change of Muscle tone | baseline: before intervention, 1st examination: finish the intervention(repetitiveTMS:10 times treatments(2weeks)；robotic GT:20 times treatments (4weeks)), 2nd examination: 7 weeks after intervention
  measure the muscle tone (kg/m) under muscle resting. Target muscles are quadriceps, hamstrings, anterior tibialis, gastrocnemius.

CONTACTS AND LOCATIONS:
Overall Officials: Ta-Sen Wei, Doctor, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No
only for research

REFERENCES:
- [Background] Brunt D, Greenberg B, Wankadia S, Trimble MA, Shechtman O. The effect of foot placement on sit to stand in healthy young subjects and patients with hemiplegia. Arch Phys Med Rehabil. 2002 Jul;83(7):924-9. doi: 10.1053/apmr.2002.3324. PMID 12098151
- [Background] Dettmann MA, Linder MT, Sepic SB. Relationships among walking performance, postural stability, and functional assessments of the hemiplegic patient. Am J Phys Med. 1987 Apr;66(2):77-90. PMID 3578493
- [Background] Hidler J, Nichols D, Pelliccio M, Brady K. Advances in the understanding and treatment of stroke impairment using robotic devices. Top Stroke Rehabil. 2005 Spring;12(2):22-35. doi: 10.1310/RYT5-62N4-CTVX-8JTE. PMID 15940582
- [Background] Kakuda W, Abo M, Watanabe S, Momosaki R, Hashimoto G, Nakayama Y, Kiyama A, Yoshida H. High-frequency rTMS applied over bilateral leg motor areas combined with mobility training for gait disturbance after stroke: a preliminary study. Brain Inj. 2013;27(9):1080-6. doi: 10.3109/02699052.2013.794973. PMID 23834634
- [Background] Kim J, Park JH, Yim J. Effects of respiratory muscle and endurance training using an individualized training device on the pulmonary function and exercise capacity in stroke patients. Med Sci Monit. 2014 Dec 5;20:2543-9. doi: 10.12659/MSM.891112. PMID 25488849
- [Background] Hornby TG, Campbell DD, Kahn JH, Demott T, Moore JL, Roth HR. Enhanced gait-related improvements after therapist- versus robotic-assisted locomotor training in subjects with chronic stroke: a randomized controlled study. Stroke. 2008 Jun;39(6):1786-92. doi: 10.1161/STROKEAHA.107.504779. Epub 2008 May 8. PMID 18467648
- [Background] Israel JF, Campbell DD, Kahn JH, Hornby TG. Metabolic costs and muscle activity patterns during robotic- and therapist-assisted treadmill walking in individuals with incomplete spinal cord injury. Phys Ther. 2006 Nov;86(11):1466-78. doi: 10.2522/ptj.20050266. PMID 17079746
- [Background] Kim P, Warren S, Madill H, Hadley M. Quality of life of stroke survivors. Qual Life Res. 1999 Jun;8(4):293-301. doi: 10.1023/a:1008927431300. PMID 10472161
- [Background] Macko RF, Ivey FM, Forrester LW, Hanley D, Sorkin JD, Katzel LI, Silver KH, Goldberg AP. Treadmill exercise rehabilitation improves ambulatory function and cardiovascular fitness in patients with chronic stroke: a randomized, controlled trial. Stroke. 2005 Oct;36(10):2206-11. doi: 10.1161/01.STR.0000181076.91805.89. Epub 2005 Sep 8. PMID 16151035
- [Background] Ng SS, Hui-Chan CW. The timed up & go test: its reliability and association with lower-limb impairments and locomotor capacities in people with chronic stroke. Arch Phys Med Rehabil. 2005 Aug;86(8):1641-7. doi: 10.1016/j.apmr.2005.01.011. PMID 16084820
- [Background] Nichols DS. Balance retraining after stroke using force platform biofeedback. Phys Ther. 1997 May;77(5):553-8. doi: 10.1093/ptj/77.5.553. PMID 9149764
- [Background] Wang RY, Tseng HY, Liao KK, Wang CJ, Lai KL, Yang YR. rTMS combined with task-oriented training to improve symmetry of interhemispheric corticomotor excitability and gait performance after stroke: a randomized trial. Neurorehabil Neural Repair. 2012 Mar-Apr;26(3):222-30. doi: 10.1177/1545968311423265. Epub 2011 Oct 5. PMID 21974983